CLINICAL TRIAL: NCT02883153
Title: Zirconium-89-girentuximab PET/CT Imaging in Patients Suspected of Primary or Relapse Clear Cell Renal Cell Carcinoma: The Impact on Clinical Decision Making.
Brief Title: Zirconium-89-girentuximab PET/CT Imaging in Renal Cell Carcinoma
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 08121986
Record Dates: First submitted 2016-08-25; First posted 2016-08-30 (Estimated); Last update posted 2017-06-19 (Actual); Status verified 2017-06

CONDITIONS: Renal Cell Carcinoma
Keywords: Zirconium-89; PET/CT; imaging; girentuximab
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — G250 monoclonal antibody

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Zirconium-89 girentuximab PET/CT (Experimental): A Zirconium-89-girentuximab PET/CT will be performed 4-5 days after single intravenous injection of 5 mg Zirconium-89-girentuximab (37 MBq).
  Interventions: Drug: Zirconium-89 girentuximab PET/CT

INTERVENTIONS:
Drug: Zirconium-89 girentuximab PET/CT — Thirty patients (suspected of ccRCC) will be included in whom conventional diagnostics are inconclusive. During a multidisciplinary team (MDT) the hypothetical next step in the clinical process will be noted. Subsequently, in these patients a Zirconium-89-girentuximab PET/CT will be performed 4-5 days after single intravenous injection of 5 mg Zirconium-89-girentuximab (37 MBq). The results of the PET/CT will be discussed during the MDT and will be used to decide what the next step in the clinical process will be. This step will be compared with the hypothetical next step from the MDT before the scan. Whether or not the PET/CT scan had impact on clinical decision making will be assessed for each individual patient.
  Other Names: girentuximab

SUMMARY:
Girentuximab is an antibody against Carbonic Anhydrase IX (CAIX), an antigen that is expressed on the cell surface of 95% of clear cell RCC (ccRCC). Zr-89-girentuximab PET/CT (Positron Emission Tomography) may be a valuable imaging technique in the diagnosis of patients with RCC. The aim of the present study is to show the impact of the Zr-89-girentuximab PET/CT on the clinical management of ccRCC patients.

DETAILED DESCRIPTION:
More advanced imaging methods are needed to reliably distinguish benign small renal masses (SRM) from renal cell carcinoma (RCC) to prevent invasive biopsies or unnecessary surgery. Similarly, improved imaging methods are needed for unambiguous detection of lesions suspect for metastatic and relapse RCC during follow-up. Girentuximab is an antibody against Carbonic Anhydrase IX (CAIX), an antigen that is expressed on the cell surface of 95% of clear cell RCC (ccRCC). Zr-89-girentuximab PET/CT may be a valuable imaging technique in the diagnosis of patients with RCC. The aim of the present study is to show the impact of the Zr-89-girentuximab PET/CT on the clinical management of ccRCC patients. Thirty patients will be included in whom conventional diagnostics are inconclusive. During a multidisciplinary team (MDT) the hypothetical next step in the clinical process will be noted (e.g. further diagnostics, treatment or active surveillance). Subsequently, in these patients a Zirconium-89-girentuximab PET/CT will be performed. Patients will receive a single intravenous dose of 5 mg Zirconium-89-girentuximab (37 MBq). A PET/CT scan will be acquired 4 or 5 days after injection. The Zirconium-89-girentuximab PET/CT will be read by a clinician with extensive experience in radiolabeled girentuximab imaging. The results of the PET/CT will be discussed during the MDT and will be used to decide what the next step in the clinical process will be. This step will be compared with the hypothetical next step from the MDT before the scan.

ELIGIBILITY:
Inclusion Criteria:

In order to participate in this study, a subject must meet all of the following criteria:

1. His or her clinician should face a diagnostic dilemma; e.g.

   * patients with a renal mass of unknown origin, or
   * patients with a primary renal mass in whom it is unclear whether there is metastatic disease, or
   * patients with a history of clear cell RCC with a suspicion of relapse or metastatic disease.
2. Minimum age 18 years
3. Signed informed consent

Exclusion Criteria:

* History of a CAIX-negative or non clear cell RCC.
* Administration of tyrosine kinase inhibiters within 1 month prior to inclusion.
* Any medical condition present that in the opinion of the investigator will affect patients' clinical status. - Administration of a radioisotope within 10 physical half lives prior to study enrollment
* Pregnancy or lactation.
* Known hypersensitivity or HACA (human anti chimeric antibodies) against Girentuximab.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2017-06-06 (Actual); Study Completion 2017-06-06 (Actual)

PRIMARY OUTCOMES:
Impact on clinical decision making | 1 year
  Impact on clinical decision making, defined as present or absent:
  * Absent: e.g. no change in treatment or follow-up
  * Present: e.g. change in follow-up schedule, change in surgical technique, change from surgery to active surveillance, or change from surgery to systemic treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Wim JG Oyen, MD, Principal Investigator — Radboud University Medical Center; Peter FA Mulders, MD, Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboudumc, Nijmegen, Netherlands

IPD SHARING:
Plan to Share IPD: No
Data will be published anonymously